CLINICAL TRIAL: NCT03249233
Title: Changes in Corneal Thickness in Keratoconic Eyes With Variation in Scleral Contact Lens Central Clearance
Brief Title: Corneal Thickness Changes With Scleral Contact Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Waterloo (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Luigina Sorbara, Associate Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22186
Record Dates: First submitted 2017-06-15; First posted 2017-08-15 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Keratoconus; Healthy Controls
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Keratoconics wearing ZenLens with high central clearance (Experimental): Scleral contact lenses designed to provide approximately 450 microns of central clearance.
  Interventions: Device: ZenLens™
- Keratoconics wearing ZenLens with low central clearance (Experimental): Scleral contact lenses designed to provide approximately 350 microns of central clearance.
  Interventions: Device: ZenLens™
- Healthy controls wearing ZenLens with high central clearance (Active Comparator): Scleral contact lenses designed to provide approximately 450 microns of central clearance.
  Interventions: Device: Zen™ RC
- Healthy controls wearing ZenLens with low central clearance (Active Comparator): Scleral contact lenses designed to provide approximately 350 microns of central clearance.
  Interventions: Device: Zen™ RC

INTERVENTIONS:
Device: ZenLens™ — The ZenLens™ semi-scleral lenses are manufactured by Alden Optic Laboratories Inc., Lancaster, NY. They will be made in Boston XO material.
  Arms: Keratoconics wearing ZenLens with high central clearance; Keratoconics wearing ZenLens with low central clearance
Device: Zen™ RC — The Zen™ RC semi-scleral lenses are manufactured by Alden Optic Laboratories Inc., Lancaster, NY. They will be made in Boston XO material.
  Arms: Healthy controls wearing ZenLens with high central clearance; Healthy controls wearing ZenLens with low central clearance

SUMMARY:
The purpose of this study is to investigate changes in the corneal thickness of scleral contact lens wearers in a keratoconic (KC) population and compare to age-matched controls. The hypothesis is that scleral contact lens wear is associated with low levels of corneal hypoxia including measurable changes in corneal thickness. Corneal thickness will be altered post scleral lens wear compared to pre-lens wear and the amount of alteration will correlate to the fitting characteristics in the central zone of the scleral lenses. We propose to take a sample of keratoconic and control participants, fit them in scleral lenses, and to measure topographic corneal thickness after 8-10 hours of scleral lens wear after three weeks of wear, to compare two instruments in the measurement of corneal thickness, and to compare the effects of varying central corneal clearance of the scleral lens on corneal thickness.

DETAILED DESCRIPTION:
The purpose of this study is to investigate changes in the corneal thickness of scleral contact lens wearers in a keratoconic (KC) population and compare to age-matched controls. The hypothesis is that scleral contact lens wear is associated with low levels of corneal hypoxia including measurable changes in corneal thickness.

This will be a prospective, dispensing study design. The study will involve up to 20 keratoconic participants and up to 20 age matched controls. Participants will attend 1 screening/fitting visit wearing their habitual contact lenses where the two test lens designs (350 and 450microns) will be fitted. There will then be a delivery visit for each design (randomly selected) and a single follow up visit after 8-10 hours of scleral lens wear, three weeks later. A washout period of a minimum of 48 hours will be applied between the cross-over of each lens design. Lenses to be worn in this study will be made of Boston XO material and are approved by Health Canada. The lenses will have a diameter of 14.8-17.0mm with a high and low sagittal depth in the corneal zone. As to which of the two lenses is being assessed, both the investigator and the participant will be masked as the assistant will provide the lenses in an unlabeled case. Masking the investigator will prevent bias when measuring corneal thickness and analyzing the data. The objectives of this study are to take a sample of keratoconic and control participants, fit them in scleral lenses, and to measure topographic corneal thickness after 8-10 hours of scleral lens wear after three weeks of wear, to compare two instruments in the measurement of corneal thickness, and to compare the effects of varying central corneal clearance of the scleral lens on corneal thickness. Secondary objectives include comparing ocular physiological outcomes between the two test lens designs. Corneal thickness will be altered post scleral lens wear compared to pre-lens wear and the amount of alteration will correlate to the fitting characteristics in the central zone of the scleral lenses.

ELIGIBILITY:
Inclusion Criteria (Test Group):

* Had been diagnosed with keratoconus in at least one eye.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.

Inclusion Criteria (Control Group)

* Had been NOT diagnosed with keratoconus in at least one eye.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.

Exclusion Criteria (Test Group):

* Is using any topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities and active neovascularization.
* Is aphakic.
* Has undergone penetrating keratoplasty.
* Is participating in any other type of eye related clinical or research study.
* Has any known allergies or sensitivity to the diagnostic pharmaceuticals or products, such as fluorescein, used in this study.

Exclusion Criteria (Control Group):

* Is using any topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities and active neovascularization.
* Is aphakic.
* Has undergone any corneal surgery.
* Is participating in any other type of eye related clinical or research study.
* Has any known allergies or sensitivity to the diagnostic pharmaceuticals or products, such as fluorescein, used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Corneal Thickness | 6 weeks
  Corneal thickness after 8-10 hours of scleral contact lens wear will be measured with the Spectralis OCT and Oculus Pentacam

SECONDARY OUTCOMES:
Visual acuity | 6 weeks
  Both high and low contrast visual acuity will be measured before and after 8-10 hours of scleral contact lens wear
Conjunctival redness | 6 weeks
  Conjunctival redness will be measured with the Keratograph before and after 8-10 hours of scleral lens wear
Corneal and conjunctival staining | 6 weeks
  Corneal and conjunctival staining will be assessed with the Keratograph and biomicroscope before and after 8-10 hours of scleral lens wear
Tear biochemistry: proteases and cytokines | 6 weeks
  The level of proteases (MMP-1, MMP-9) and cytokines (IL-1, IL-6, IL-8, TNFα) in each of the tear samples collected from the lenses will be measured using the Meso Scale Discovery System (MSD-ECL) before and after 8-10 hours of scleral lens wear.
Tear biochemistry: cell count | 6 weeks
  Polymorphonuclear leukocyte (PMN) cells in each of the tear samples collected from the lenses will be analyzed and counted using the BD FACS Calibur™ Flow Cytometer and Bright-Line Hemacytometer before and after 8-10 hours of scleral lens wear.

CONTACTS AND LOCATIONS:
Overall Officials: Luigina Sorbara, OD MSc, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo School of Optometry and Vision Science, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Worp E, Bornman D, Ferreira DL, Faria-Ribeiro M, Garcia-Porta N, Gonzalez-Meijome JM. Modern scleral contact lenses: A review. Cont Lens Anterior Eye. 2014 Aug;37(4):240-50. doi: 10.1016/j.clae.2014.02.002. Epub 2014 Mar 12. PMID 24631015
- [Background] Romero-Rangel T, Stavrou P, Cotter J, Rosenthal P, Baltatzis S, Foster CS. Gas-permeable scleral contact lens therapy in ocular surface disease. Am J Ophthalmol. 2000 Jul;130(1):25-32. doi: 10.1016/s0002-9394(00)00378-0. PMID 11004256
- [Background] Walker MK, Bergmanson JP, Miller WL, Marsack JD, Johnson LA. Complications and fitting challenges associated with scleral contact lenses: A review. Cont Lens Anterior Eye. 2016 Apr;39(2):88-96. doi: 10.1016/j.clae.2015.08.003. Epub 2015 Sep 2. PMID 26341076
- [Background] Ucakhan OO, Ozkan M, Kanpolat A. Corneal thickness measurements in normal and keratoconic eyes: Pentacam comprehensive eye scanner versus noncontact specular microscopy and ultrasound pachymetry. J Cataract Refract Surg. 2006 Jun;32(6):970-7. doi: 10.1016/j.jcrs.2006.02.037. PMID 16814055
- [Background] Liesegang TJ. Contact lens-related microbial keratitis: Part I: Epidemiology. Cornea. 1997 Mar;16(2):125-31. PMID 9071523